CLINICAL TRIAL: NCT02730208
Title: A Phase 2, Randomized, Placebo-Controlled, Double-blind Study to Evaluate the Effect of VX-661 in Combination With Ivacaftor on Chest Imaging Endpoints in Subjects Aged 12 Years and Older With Cystic Fibrosis, Homozygous for the F508del CFTR Mutation
Brief Title: A Study to Evaluate the Effect of VX-661 in Combination With Ivacaftor on Chest Imaging Endpoints in Subjects With Cystic Fibrosis, Homozygous for the F508del CFTR Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX15-661-112
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEZ/IVA (Experimental): Participants received TEZ 100 milligram (mg)/IVA 150 mg fixed dose combination tablet orally once daily in the morning and IVA 150 mg tablet orally once daily in the evening for 72 weeks.
  Interventions: Drug: Tezacaftor/Ivacaftor; Drug: Ivacaftor
- Placebo (Placebo Comparator): Participants received placebo matched to TEZ/IVA fixed dose combination tablet orally once daily in the morning and placebo matched to IVA tablet orally once daily in the evening for 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tezacaftor/Ivacaftor — TEZ 100 mg/IVA 150 mg fixed-dose combination tablet.
  Other Names: TEZ/IVA; VX-661/VX-770
  Arms: TEZ/IVA
Drug: Ivacaftor — IVA 150 mg tablet.
  Other Names: VX-770; IVA
  Arms: TEZ/IVA
Drug: Placebo — Placebo matched to TEZ/IVA fixed-dose combination tablet.
  Arms: Placebo
Drug: Placebo — Placebo matched to IVA tablet.
  Arms: Placebo

SUMMARY:
The primary purpose of study is to evaluate the treatment effect of tezacaftor in combination with ivacaftor (TEZ/IVA) on chest imaging endpoints using low-dose computed tomography (LDCT) at Week 72, and to evaluate the safety of TEZ/IVA through Week 72.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous for the F508del CFTR mutation
* Confirmed diagnosis of CF
* Percent predicted forced expiratory volume (ppFEV1) ≥70% of predicted normal for age, sex, and height during screening.
* Stable CF disease as judged by the investigator

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 28 days before Day 1 (first dose of study drug)
* Pregnant or nursing females.
* Sexually active subjects of reproductive potential who are not willing to follow the contraception requirements.
* Any contraindication to undergoing chest imaging, as per the site's institutional guidelines

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Australia (9):
  - Chermside
  - Melbourne
  - Nedlands
  - New Lambton Heights
  - Parkville SIC
  - Randwick
  - South Brisbane
  - Subiaco
  - Westmead

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 41 participants were randomized and treated in the study.
Period: Overall Study
Arm/Group | TEZ/IVA | Placebo
Started | 20 | 21
Completed | 20 | 20
Not Completed | 0 | 1
Not completed — Withdrawal of consent (not due to AE) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TEZ/IVA: Participants received TEZ 100 mg/IVA 150 mg fixed dose combination tablet orally once daily in the morning and IVA 150 mg tablet orally once daily in the evening for 72 weeks.
- Total: Total of all reporting groups
Arm/Group | TEZ/IVA | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.4 (7.5) | 20.1 (9.3) | 20.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Total Brody/Cystic Fibrosis - Computed Tomography (CF-CT) Score [Mean (Standard Deviation); unit: scores on a scale] — The exploratory Brody/CF-CT score semi-quantitatively scores the degree of structural lung disease as shown on CT in participants with CF. The score ranges from a minimum of 0 to a maximum of 219 with higher scores indicating more severe structural lung disease.
  scores on a scale | 38.29 (22.91) | 43.68 (33.96) | 40.98 (28.72)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Total Brody/CF-CT Score
Description: The exploratory Brody/CF-CT score semi-quantitatively scores the degree of structural lung disease as shown on CT in participants with CF. The score ranges from a minimum of 0 to a maximum of 219 with higher scores indicating more severe structural lung disease.
Time Frame: From Baseline at Week 72
Population: FAS included all participants who were randomized and received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | TEZ/IVA | Placebo
Number analyzed (Participants) | 20 | 21
scores on a scale | 0.90 (2.09) | 2.38 (2.07)
Statistical Analysis 1: Comparison: TEZ/IVA vs Placebo; Test type: Other — Treatment effect outcomes are estimates; Least Squares (LS) Mean Difference = -1.48, 95% CI 2-sided [-7.47 to 4.52]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 76
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TEZ/IVA | Placebo
Number analyzed (Participants) | 20 | 21
Participants
  Participants with AEs | 20 | 21
  Participants with SAEs | 8 | 13

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 76
Arm/Group | TEZ/IVA | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 8/20 | 13/21
Other Adverse Events (participants affected / at risk) | 19/20 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEZ/IVA (N=20) | Placebo (N=21)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 5 | 6
Lung infection pseudomonal (Infections and infestations) | 2 | 0
Atypical mycobacterial lower respiratory tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Type I hypersensitivity (Immune system disorders) | 0 | 1
Bacterial test positive (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TEZ/IVA (N=20) | Placebo (N=21)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 5 | 9
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Lower respiratory tract infection bacterial (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pyrexia (General disorders) | 3 | 2
Fatigue (General disorders) | 1 | 2
Chest pain (General disorders) | 0 | 2
Migraine (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 3
Sunburn (Injury, poisoning and procedural complications) | 1 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2
Fungal test positive (Investigations) | 1 | 2
Bacterial test positive (Investigations) | 0 | 5
Blood alkaline phosphatase increased (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT02730208/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT02730208/SAP_001.pdf